CLINICAL TRIAL: NCT03763409
Title: The Effect of Losartan on Emotional Memory in Healthy Volunteers
Brief Title: Losartan and Emotional Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R56384/RE001
Record Dates: First submitted 2018-11-27; First posted 2018-12-04 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Memory; Learning
Keywords: anxiety; losartan; appetitive learning; aversive learning
MeSH Terms: conditions — Anxiety Disorders | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: Parallel randomised
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- losartan (Experimental): 50 mg single-dose oral losartan
  Interventions: Drug: Losartan Potassium
- placebo (Placebo Comparator): microcellulose placebo in identical capsule
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Losartan Potassium — active drug
  Arms: losartan
Other: placebo — placebo
  Arms: placebo

SUMMARY:
This study explores the effects of single-dose losartan (50mg) versus identical placebo capsule on emotional memory and learning in healthy volunteers.

DETAILED DESCRIPTION:
The commonly prescribed antihypertensive drug losartan (brand name: Cozaar; UK licensed for 20 years) targets the renin-angiotensin system - a hormone system regulating blood pressure - by acting as an angiotensin receptor antagonist. In particular, the drug prevents a docking of the protein angiotensin IV to AT1 receptors, which leads to a dilation if vessels and a reduction in blood pressure. However, the increase in free angiotensin IV has also been associated with an increase in synaptic plasticity, the cellular mechanism involved in learning and memory. As such, losartan appears to have cognition-enhancing properties, in a way that a single dose of 50mg improves prospective memory in healthy humans. However, preliminary pre-clinical results also suggest that a single injection of the drug improves fear extinction in rodents, which is the equivalent to human cognitive-behavioural therapy for anxiety disorders. Furthermore, compared to other antihypertensive drugs, regular losartan treatment appears to prevent the development of post-traumatic stress disorder symptoms following trauma exposition. Such results suggest that the renin-angiotensin system plays a key role in the development and extinction of anxiety, and that adding losartan to cognitive-behavioural therapy for anxiety in humans might have synergistic effects. However, it remains to be clarified what the basic effects of this drug on emotional information processing in humans are to identify mechanisms by which it may improve psychological treatments.

In this study, the key neuropsychological effects of probing the renin-angiotensin system on emotional information processing and learning will be investigated. In a double-blind, randomised between-groups design, 54 healthy volunteers will be randomised to a group receiving a single dose of losartan (50mg) versus placebo. When peak plasma levels are reached, participants will work on a battery of behavioural measures of emotional information processing and learning.

The results from this study will help understand how the renin-angiotensin system affects emotional information processing and learning, and they will help establish a battery of tasks that sensitively respond to such manipulations. Such information will ultimately lead to the development of losartan and similar agents for the more effective and more compact treatment of anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to provide informed consent
* male or Female, aged 18-50
* body mass index (BMI) of 18-30 kg/m2
* fluent English skills
* non- or light-smoker (< 5 cigarettes a day)

Exclusion Criteria:

* Female participant who is pregnant or breast-feeding
* CNS-active medication during the last 6 weeks
* Current blood pressure or other heart medication (especially aliskiren or beta blockers)
* Intravascular fluid depletion
* Past or present DSM-IV axis-I diagnosis or suspected diagnosis (from SCID results at screening)
* Alcohol or substance abuse
* First-degree family member with a history of a severe psychiatric disease
* Impaired liver or kidney function
* Lifetime history of epilepsy or other neurological disease, systemic infection, or clinically significant hepatic, cardiac, obstructive respiratory, renal, cerebrovascular, metabolic, endocrine or pulmonary disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Insufficient English skills
* participated in another study involving CNS-active medication during the last 6 weeks

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
aversive and appetitive learning | 1 hour after capsule intake
  a learning task wil assess to what degree participants learn from win versus loss outcomes in different environments

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pulcu E, Shkreli L, Holst CG, Woud ML, Craske MG, Browning M, Reinecke A. The Effects of the Angiotensin II Receptor Antagonist Losartan on Appetitive Versus Aversive Learning: A Randomized Controlled Trial. Biol Psychiatry. 2019 Sep 1;86(5):397-404. doi: 10.1016/j.biopsych.2019.04.010. Epub 2019 Apr 17. PMID 31155138